CLINICAL TRIAL: NCT00973583
Title: Vitamin D Supplementation for the Prevention of Acute Respiratory Tract Infections; a Randomized Double-blinded Trial in Young Finnish Men
Brief Title: Vitamin D Supplementation for the Prevention of Acute Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Finnish Defense Forces (Other Government)
Responsible Party: Principal Investigator, Ilkka Laaksi, M.D. PhD, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UTampere-RO5125
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Respiratory Tract Infections
Keywords: vitamin D; infection; Vitamin D for the prevention of respiratory tract infections
MeSH Terms: conditions — Respiratory Tract Infections; Infections | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D (Active Comparator)
  Interventions: Dietary Supplement: vitamin D
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: vitamin D — vitamin D3 400 IU daily
  Other Names: Minisun
  Arms: vitamin D
Dietary Supplement: placebo — placebo
  Other Names: Pharmia, Finland
  Arms: placebo

SUMMARY:
The investigators earlier clinical study in 754 young Finnish men demonstrated a significant negative association of serum 25-OHD concentration with acute respiratory tract infections. The present study aimed to determine whether vitamin D supplementation may decrease the incidence of acute respiratory tract infections.

DETAILED DESCRIPTION:
Subjects comprised 164 male conscripts at a military base in Finland. Half of the participants were randomly allocated to receive 400 IU vitamin D daily and half received placebo from October through March. Serum vitamin D and plasma parathyroid hormone concentrations were determined. Subjects were followed for 6 months and the primary outcome was the number of days absent from duty due to ARTI.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Use vitamin D

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2005-05; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of days absent from duty due to respiratory tract infection | 6 months

SECONDARY OUTCOMES:
The proportion of men remaining healthy throughout the 6-month study period | 6 months
The number needed to treat calculated from the proportion of men without any days absent from duty | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka T Laaksi, M.D., Principal Investigator — Tampere University; Harri Pihlajamaki, Docent, Study Director — Research Department, Centre for Military Medicine, Helsinki, Finland
Locations (1):
- university of Tampere, Tampere, Finland